CLINICAL TRIAL: NCT02518230
Title: Respiratory Severity and Caloric Consumption on NAVA: Randomized Crossover Trial of NAVA and SIMV
Brief Title: Randomized Crossover of NAVA and Synchronized Intermittent Pressure Ventilation in Neonates and Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Crossover NAVA
Record Dates: First submitted 2015-08-03; First posted 2015-08-07 (Estimated); Results first posted 2021-07-23 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-06

CONDITIONS: Respiratory Insufficiency; Infant, Newborn, Disease
MeSH Terms: conditions — Respiratory Insufficiency; Disease | interventions — Interactive Ventilatory Support

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neurally Adjusted Ventilatory Assist (Other): Subject will be randomized to NAVA ventilation. Intervention is mechanical ventilation with Neurally Adjusted Ventilatory Assist for 12 hours.
  Interventions: Device: Neurally Adjusted Ventilatory Assist; Device: Synchronized Interm. Mandatory Assist
- Synchronized Interm. Mandatory Assist (Other): Subject will be randomized to SIMV(PC)PS ventilation. Intervention is mechanical ventilation with Synchronized Intermittent Mandatory Assist with Pressure Support for 12 hours.
  Interventions: Device: Neurally Adjusted Ventilatory Assist; Device: Synchronized Interm. Mandatory Assist

INTERVENTIONS:
Device: Neurally Adjusted Ventilatory Assist — The subject will be crossed over from the baseline ventilator mode to Neurally Adjusted Ventilatory Assist
Device: Synchronized Interm. Mandatory Assist — The subject will be crossed over from the baseline ventilator mode to Synchronized Intermittent Mandatory Assist with Pressure Support

SUMMARY:
This study is a single center, prospective cohort crossover study comparing mechanically ventilated neonates and infants on Neurally Adjusted Ventilatory Assist (NAVA) and synchronized intermittent mandatory ventilation with pressure control plus pressure support (SIMV(PC) + PS) modes.

This design will allow for direct comparison of two commonly used ventilator modalities in the neonatal intensive care unit (NICU) to determine if one mode is superior to the other with regards to respiratory mechanics and estimated energy expenditure.

It is hypothesized that neonates and infants will have improved respiratory severity score (MAP X FiO2) utilizing NAVA compared to the SIMV (PC) + PS mode but will have increased estimated energy expenditure.

DETAILED DESCRIPTION:
This single center, prospective cohort crossover study will involve mechanically ventilated neonates and infants who are determined to be on stable ventilator settings in either the NAVA or SIMV(PC) + PS modes. This design will allow for direct comparison of two commonly used ventilator modalities in the neonatal intensive care unit (NICU) to determine if one mode is superior to the other with regards to respiratory mechanics and energy expenditure.

Infants will be screened for stability criteria including: being stable on the ventilator in either SIMV (PC) + PS or NAVA mode, on weaning or unchanged ventilatory support in previous 12 hours, and no need of escalation of ventilatory pressure or rate in prior 12 hours.

After screening criteria is met and consent has been obtained, data will be retrospectively collected for 12 hours prior to randomization. After the subject is randomized, the infant will be stabilized and data will be collected for 12 hours in the randomized mode. Data will then be collected for 12 hours afterwards in the crossover mode. Data will be collected in areas of patient demographics, diagnoses, indications for mechanical ventilation, hemodynamic variables and respiratory parameters. While in each mode, the patient will also have indirect calorimetry obtained to determine estimated energy expenditure of each mode.

ELIGIBILITY:
Inclusion Criteria:

* Neonates and infants, 22 weeks gestation age or older at birth
* Require mechanical ventilation for respiratory support in either SIMV (PC) + PS or NAVA modes
* Stable on the ventilator with a fractional inspired oxygen requirement (FiO2) of 0.60 or less.
* Stable on the ventilator with weaning or unchanged ventilatory support without need of escalation of ventilatory pressure or rate in prior 12 hours.

Exclusion Criteria:

* Major congenital anomalies
* Neurologic compromise of respiratory drive
* Phrenic nerve palsy
* Sedated enough to suppress respiratory drive
* Respiratory support with volume mechanical ventilation
* Respiratory support with high frequency oscillatory ventilation

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jamie L Rosterman, DO, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

REFERENCES:
- [Derived] Rosterman JL, Pallotto EK, Truog WE, Escobar H, Meinert KA, Holmes A, Dai H, Manimtim WM. The impact of neurally adjusted ventilatory assist mode on respiratory severity score and energy expenditure in infants: a randomized crossover trial. J Perinatol. 2018 Jan;38(1):59-63. doi: 10.1038/jp.2017.154. Epub 2017 Oct 26. PMID 29072677

RESULTS

PARTICIPANT FLOW:
Groups:
- NAVA Ventilation First, Then SIMV(PC)PS Ventilation: Subject will be randomized to NAVA ventilation first. Intervention is mechanical ventilation with Neurally Adjusted Ventilatory Assist for 12 hours. Subjects will cross over.
  Neurally Adjusted Ventilatory Assist: The subject will be crossed over from the baseline ventilator mode to Neurally Adjusted Ventilatory Assist
  Synchronized Interm. Mandatory Assist: The subject will be crossed over from the baseline ventilator mode to Synchronized Intermittent Mandatory Assist with Pressure Support
- SIMV(PC)PS Ventilation First, Then NAVA Ventilation: Subject will be randomized to SIMV(PC)PS ventilation first. Intervention is mechanical ventilation with Synchronized Intermittent Mandatory Assist with Pressure Support for 12 hours. Subjects will cross over
  Neurally Adjusted Ventilatory Assist: The subject will be crossed over from the baseline ventilator mode to Neurally Adjusted Ventilatory Assist
  Synchronized Interm. Mandatory Assist: The subject will be crossed over from the baseline ventilator mode to Synchronized Intermittent Mandatory Assist with Pressure Support
Period: Overall Study
Arm/Group | NAVA Ventilation First, Then SIMV(PC)PS Ventilation | SIMV(PC)PS Ventilation First, Then NAVA Ventilation
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SIMV(PC)PS Ventilation First, Then NAVA Ventilation: Subject will be randomized to SIMV(PC)PS ventilation first. Intervention is mechanical ventilation with Synchronized Intermittent Mandatory Assist with Pressure Support for 12 hours. subjects will cross over.
  Neurally Adjusted Ventilatory Assist: The subject will be crossed over from the baseline ventilator mode to Neurally Adjusted Ventilatory Assist
  Synchronized Interm. Mandatory Assist: The subject will be crossed over from the baseline ventilator mode to Synchronized Intermittent Mandatory Assist with Pressure Support
- Total: Total of all reporting groups
Arm/Group | NAVA Ventilation First, Then SIMV(PC)PS Ventilation | SIMV(PC)PS Ventilation First, Then NAVA Ventilation | Total
Number analyzed (Participants) | 11 | 11 | 22
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 11 | 22
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Full Range); unit: Post Menstral Age in weeks] | 32 [28 to 44] | 32 [28 to 44] | 32 [28 to 44]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 6 | 7 | 13
Region of Enrollment [Number; unit: participants]
  United States | 11 | 11 | 22

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Severity Score (MAP X FiO2)
Description: The respiratory severity score will be calculated throughout 24 hour time frame prior to and after study initiation to determine the subject's respiratory severity prior to the randomization, after randomization and after crossover. The respiratory severity score (RSS) is a simplified severity score consisting of the mean airway pressure (MAP) multiplied by the fraction of inspired oxygen (FiO2). This score ranges from 0 to 12, with a higher score indicating more severe disease.
Time Frame: 12 hours and 24 hours
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- NAVA Ventilation First, Then SIMV(PC)PS Ventilation: Intervention is mechanical ventilation with Neurally Adjusted Ventilatory Assist for 12 hours.
- SIMV(PC)PS Ventilation First, Then NAVA Ventilation: Intervention is mechanical ventilation with Synchronized Intermittent Mandatory Assist with Pressure Support for 12 hours.
Arm/Group | NAVA Ventilation First, Then SIMV(PC)PS Ventilation | SIMV(PC)PS Ventilation First, Then NAVA Ventilation
Number analyzed (Participants) | 11 | 11
score on a scale
  Respiratory severity score 12 h average | 3.83 (2) | 3.82 (1.79)
  Respiratory severity score 24 h average | 3.46 (2.24) | 3.86 (1.93)

2. Secondary Outcome: Energy Expenditure
Description: The subject will have indirect calorimetry performed twice during the study on each mode, 12 hours after randomization and 12 hours after crossover to determine the approximate amount of energy expenditure needed for each mode of mechanical ventilation.
  Energy expenditure is calculated by using the Harris-Benedict equation, resulted in kcal/kg per day.
Time Frame: 12 hours and 24 hours
Population: This outcome measure was not broken down by intervention as it is a median of energy expenditure for all participants enrolled. The data herein are cumulative for all study participants.
Measure: Median (Inter-Quartile Range); unit: kcal/kg per day
Groups:
- Overall Study: Overall Study, Outcome not broken down further
Arm/Group | Overall Study
Number analyzed (Participants) | 22
kcal/kg per day | 25.6 [16.1 to 46.5]

ADVERSE EVENTS:
Time Frame: 24 hours
Description: Escalation of ventilation settings
Arm/Group | NAVA Ventilation First, Then SIMV(PC)PS Ventilation | SIMV(PC)PS Ventilation First, Then NAVA Ventilation
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/11
Other Adverse Events (participants affected / at risk) | 0/11 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes